CLINICAL TRIAL: NCT06041217
Title: Efficacy and Safety of Semaglutide 2.4 mg Once-weekly in Adults With Overweight and Obesity
Brief Title: A Research Study to See How Well Semaglutide Helps People Who Have a Body Weight Above the Healthy Weight Range
Acronym: STEP12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4706; U1111-1273-4538 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide 2.4 milligram (mg) (Experimental): Participants will receive once-weekly subcutaneous (s.c) injection of semaglutide for 44 weeks.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive once-weekly subcutaneous (s.c) injection of placebo for 44 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Subcutaneous injections of semaglutide once-weekly at escalating doses every fourth week until maintenance dose of 2.4 mg of semaglutide is reached.
  Arms: Semaglutide 2.4 milligram (mg)
Drug: Placebo — Subcutaneous injections of placebo once-weekly at escalation doses manner as semaglutide every fourth week until maintenance dose of placebo matched to 2.4 mg is reached.
  Arms: Placebo

SUMMARY:
This study will look at how the investigational dose of semaglutide works in helping people with excess body weight, to lose weight. This study will compare the weight loss in people taking semaglutide to people taking "dummy" medicine (placebo). The study will last for about 1 year. The participants will have 12 visits at the clinic and 3 remote visits by phone calls with the study doctor or staff.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at the time of signing informed consent.
* Body mass index (BMI) of greater than or equal to 24 and less than 28 kilogram per square meter ( kg/m^2) with the presence of at least one weight related complication (treated or untreated): Type 2 diabetes (T2D), hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease or BMI greater than or equal to 28 and less 30 kg/m^2, with or without weight related complications at screening.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.

For participants with T2D at screening:

- Diagnosed with T2D greater than or equal to 180 days prior to the day of screening

Treated with either:

* Diet and exercise alone or with 1-3 marketed oral antidiabetic drugs (metformin, alpha glucosidase, Sulfonylureas (SU), glinides, sodium-glucose co-transporter 2 inhibitors (SGLT2i) or glitazone as a single agent or in combination) according to local label.
* Treatment with oral anti-diabetic drugs should be stable (same drug(s) or active ingredient, dose, and dosing frequency) for at least 60 days before screening
* Glycated haemoglobin (HbA1c) of less than or equal to 10.0 percent (less than or equal to 86 millimoles per mol [mmol/mol]) as measured by the central laboratory at screening.

Exclusion Criteria:

* A self-reported change in body weight greater than 5 kilograms (kg) within 90 days before screening irrespective of medical records.
* Treatment with any medication for the indication of obesity within the past 90 days before screening.
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.

For participants without T2D at screening:

- HbA1c greater than or equal to 6.5percent (48 mmol/mol) as measured by the laboratory.

For participants with T2D at screening:

* Renal impairment with estimated Glomerular Filtration Rate (eGFR) value of less than 30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation as defined by Kidney Disease Improving Global Outcomes (KDIGO) 2012 classification by the central laboratory at screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%).
Body weight reduction ≥ 5% (yes/no) | At end of treatment (week 44)
  Measured as count of participants.

SECONDARY OUTCOMES:
Body weight reduction ≥ 10% (yes/no) | At end of treatment (week 44)
  Measured as count of participants.
Change in waist circumference | From baseline (week 0) to end of treatment (week 44)
  Measured in centimeter.
Change in body weight | From baseline (week 0) to end of treatment (week 44)
  Measured in kilograms (kg).
Change in body mass index | From baseline (week 0) to end of treatment (week 44)
  Measured in kilograms per square meter (kg/m^2).
Change in waist-height ratio (WtHR) | From baseline (week 0) to end of treatment (week 44)
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 44)
  Measured in millimeters of mercury (mmHg).
Change in diastolic blood pressure | From baseline (week 0) to end of treatment (week 44)
  Measured in mmHg.
Change in total cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in ratio to baseline.
Change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in ratio to baseline.
Change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in ratio to baseline.
Change in very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 44)
  Measured in ratio to baseline.
Change in triglycerides | From baseline (week 0) to end of treatment (week 44)
  Measured in ratio to baseline.
Change in free fatty acids | From baseline (week 0) to end of treatment (week 44)
  Measured in ratio to baseline.
Change in high-sensitivity c-reactive protein (hsCRP) | From baseline (week 0) to end of treatment (week 44)
  Measured in ratio to baseline.
Change in Glycated Haemoglobin (HbA1c) (Percent [%]) | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage point.
Change in HbA1c (mmol/mol) | From baseline (week 0) to end of treatment (week 44)
  Measured in millimoles per mole (mmol/mol).
Change in fasting plasma glucose (mg/dL) | From baseline (week 0) to end of treatment (week 44)
  Measured in milligrams per deciliter (mg/dL).
Change in fasting plasma glucose (mmol/L) | From baseline (week 0) to end of treatment (week 44)
  Measured in mmol/L
Number of Treatment-emergent Adverse Events (TEAEs) | From baseline (week 0) to end of treatment (week 44)
  Measured in count of events.
Number of Serious Adverse Events (SAEs) | From baseline (week 0) to end of treatment (week 44)
  Measured in count of events.
Change in pulse | From baseline (week 0) to end of treatment (week 44)
  Measured in beats per minute (bpm).
Number of clinically significant hypoglycaemic episodes (level 2) (less than [<] 3.0 millimole per liter [mmol/L]) confirmed by blood glucose [BG] meter) | From baseline (week 0) to end of study (week 49)
  Measured in number of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (21):
- China (16):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital-Endocrinology, Fuzhou, Fujian
  - Huizhou Central People's Hospital-Endocrinology, Huizhou, Guangdong
  - Hengshui People's Hospital (Harrison International Peace Hospital)-Endocrinology, Hengshui, Hebei
  - Taihe Hospital-Endocrinology, Shiyan, Hubei
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University_Nanjing, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - The First Bethune hospital of Jilin University-Endocrinology, Changchun, Jilin
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Fifth People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - Tongren Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
- Taiwan (5):
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital_main, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com
URL: http://novonordisk-trials.com